CLINICAL TRIAL: NCT00530127
Title: A Six-month Double-blind, Randomized, Placebo-controlled Study Investigating the Safety and Tolerability of Deferiprone in Patients With Friedreich's Ataxia
Brief Title: A Study Investigating the Safety and Tolerability of Deferiprone in Patients With Friedreich's Ataxia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Dian Shaw, ApoPharma Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LA29-0207
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Deferiprone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A (Placebo Comparator): Placebo solution
  Interventions: Drug: placebo
- B (Experimental): Deferiprone oral solution 20 mg/kg/day
  Interventions: Drug: deferiprone
- C (Experimental): Deferiprone oral solution 40 mg/kg/day
  Interventions: Drug: deferiprone
- D (Placebo Comparator): Placebo solution
  Interventions: Drug: placebo
- E (Experimental): deferiprone oral solution 60 mg/kg/day
  Interventions: Drug: deferiprone

INTERVENTIONS:
Drug: placebo — Same dose and frequency as treatment
  Arms: A
Drug: deferiprone — 100 mg/mL
  Arms: B
Drug: deferiprone — 100 mg/mL
  Arms: C
Drug: placebo — Same dosage and frequency as study drug
  Arms: D
Drug: deferiprone — 100 mg/mL
  Arms: E

SUMMARY:
The primary objective of this study is to demonstrate the safety and tolerability of deferiprone in subjects with Friedreich's ataxia (FRDA).

The secondary objective is to evaluate the efficacy of deferiprone for the treatment of FRDA, as assessed by a 9-Hole Peg Test (9HPT), Timed 25-Foot Walk (T25FW), Low-Contrast Letter Acuity test (LCLA), International Cooperative Ataxia Rating Scale (ICARS), and Friedreich's Ataxia Rating Scale (FARS).

The tertiary objectives are to evaluate the effect of deferiprone on:

1. cardiac function as measured by changes in Left Ventricular Shortening Fraction (LVSF), Left Ventricular Ejection Fraction (LVEF) and Left Ventricular (LV) mass using echocardiogram (ECHO),
2. quality of life using quality-of-life surveys, and
3. functional status using Activities of Daily Living (ADL).

DETAILED DESCRIPTION:
This will be a multi-centre, double-blind, randomized, placebo-controlled clinical trial. A total of 80 patients with Friedreich's ataxia will be enrolled. Eligible patients will receive deferiprone oral solution or placebo at a total daily dose of 20 mg/kg/day, 40 mg/kg/day or 60 mg/kg/day, divided into two-daily doses for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of FRDA, with confirmed mutation (excludes point mutation) in the frataxin (FXN) gene and GAA repeats ≥ 400 on the shorter allele.
2. Males or females aged 7 to 35 years.
3. No exposure to idebenone, coenzyme Q10, vitamin C, vitamin E or other antioxidants as a supplement or as a drug therapy for a period of at least one month prior to start of treatment and during the study.
4. Neurological testing: A FARS score >20 and <85 at Screening and Baseline.
5. Female subjects of childbearing potential must have a negative pregnancy test at Baseline.
6. If the subject is a heterosexual, sexually-active male, he confirms that he and/or his female partner will use an effective method of contraception for the length of the trial and for 30 days following completion of the study or early termination.
7. Signed and witnessed written informed consent/assent, obtained prior to the first study intervention, as well as the ability to adhere to study restrictions, appointments and evaluation schedule.

Exclusion Criteria:

1. Iron deficiency defined as ferritin levels below the reference range for age- and sex-matched controls
2. Unable to complete T25FW AND with score > 5 minutes in the 9HPT. (Subjects who can complete T25FW or with a score ≤ 5 minutes in the 9HPT will be allowed to enroll if the score has not doubled compared to screening).
3. Abnormal ALT, greater than 2.0 times the upper limit of normal on two consecutive assessments.
4. Serum creatinine outside the normal reference range.
5. History or evidence of neutropenia defined by an absolute neutrophil count (ANC) < 1.5 x 109/L or thrombocytopenia defined by a platelet count <150 x 109/L.
6. Refusal to participate in screening procedures or unable to participate in screening procedures or unable to comply with the requirements of the protocol.
7. Receiving any investigational drug products or having received any investigational product within 30 days prior to enrollment into this study.
8. Subjects who have previously taken deferiprone.
9. Subjects who, in the opinion of the Investigator, represent poor medical, psychological or psychiatric risks, and for whom participation in an investigational trial would be unwise.
10. Pregnant, breastfeeding or planning to become pregnant during the study period.
11. History of malignancy.
12. History of alcohol or drug abuse.
13. Investigators, site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
14. Hypersensitivity to the active substance (deferiprone) or any of the excipients in the oral solution.
15. QT interval > 450 msec at Baseline.

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The patient's tolerance of treatment will be determined, as assessed by the occurrence of adverse events | 6 months

SECONDARY OUTCOMES:
The efficacy endpoints will be change in the score for 9-Hole Peg Test (9HPT), Timed 25-Foot Walk (T25FW), Low-Contrast Letter Acuity test (LCLA), International Cooperative Ataxia Rating Scale (ICARS), and Friedreich's Ataxia Rating Scale (FARS). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Pandolfo, M.D., Principal Investigator — Hospital Erasme, Brussels, Belgium; Arnold Munnich, M.D., Principal Investigator — Hospital Necker-Enfants Malades, Paris, France; Franco Taroni, Principal Investigator — Fondazione IRCCS Istituto Neurologico "C. Besta"; Martin Delatycki, Principal Investigator — Murdoch Children's Research Institute, Vicotria, Australia; Javier Arpa, Principal Investigator — La Fundaction Para la Investigacion Biomedica, Madrid, Spain; Mark Tarnopolsky, MD, Principal Investigator — McMaster University
Locations (6):
- Murdoch Children's Research Institute, Victoria, Australia
- Hospital Erasme, Brussels, Belgium
- McMaster University, Hamilton, Ontario, Canada
- Hospital Necker-Enfants Malades, Paris, France
- Fondazione IRCCS Istituto Neurologico "C. Besta", Milan, Italy
- La Fundacion Para la Investigacion Biomedica, Madrid, Spain